CLINICAL TRIAL: NCT03837600
Title: Sputum Labeling Utilizing Synthetic Meso-Tetra (4-Carboxyphenyl) Porphyrin (TCPP) for Detection of Lung Cancer
Status: Completed | Type: Observational
Sponsor: bioAffinity Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BA-001
Record Dates: First submitted 2019-01-31; First posted 2019-02-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
Keywords: LDCT; Sputum; High-risk Smoker; Porphyrin; Early detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Cohort: Participants who have smoked less than 5 pack-years, have quit smoking for more than 15 years and have no known lung diseases.
- High-risk Cohort: Participants who are at high risk for lung cancer including current smokers who have smoked for more than 30 pack-years and have not quit within 15 years.
- Cancer Cohort: Participants who have been diagnosed with lung cancer.

SUMMARY:
The primary objective of this study is optimization of the assay to discriminate between cancer cells and non-cancer cells in sputum samples by the performance of experiments that will determine methods to liquefy sputum, select proper fixatives and buffers, determine the efficacy of use of methyl-beta-cyclodextrin (MBCD) in sputum processing and determine the use of flow cytometry for high-throughput, and in the establishment of cell count and sputum cell populations in patient samples.

The secondary objective of this study is comparison of the characteristics of sputum from three cohorts labeled with CyPath Lung to determine differential characteristics between samples taken from Participants who are not at high risk for lung cancer, Participants at high risk for lung cancer who are free of the disease and Participants with confirmed lung cancer.

DETAILED DESCRIPTION:
A clinical study was completed to determine the clinical sensitivity and specificity of the CyPath® Early Lung Cancer Detection Assay (the "Assay") by comparing sputum specimens from three cohorts of Participants including healthy individuals, individuals at high risk for lung cancer and individuals diagnosed with lung cancer. Results were published in the Journal of Thoracic Oncology- see reference. Research now is planned to optimize the Assay as described below. Therefore, collection and analysis of sputum samples from three cohorts including healthy Participants, high risk Participants and cancer patient Participants are needed to conduct continuing research leading to optimization of the Assay.

This study will be performed at multiple study centers to collect sputum samples from three cohorts including healthy Participants who have no known lung disease, individuals at high risk for lung cancer and individuals at high risk for lung cancer who have been diagnosed with lung cancer. The sputum samples will be collected at the study site or at the Participant's home after explanation of the collection procedure by study staff. Samples will be identified with an identification number blinding the sample identity. However, the cohort classification of the sputum sample will be known by the Researcher as required to conduct the experiments. In the latter phase of the study that requires comparison of results between cohorts, researchers will be blinded to the classification of the sputum sample. Each subject's sputum specimen will be processed in accordance with individual experimental protocol at the laboratory of bioAffinity Technologies, Inc. (BA) located at the University of Texas at San Antonio 1604 main campus in San Antonio, Texas. The BA laboratory will process each sputum sample for use in optimizing the Assay. bioAffinity researchers who will be blinded as to the Participant's identity will perform the experiments that will determine methods to liquefy sputum, select proper fixatives and buffers, determine the efficacy of use of methyl-beta-cyclodextrin (MBCD) in sputum processing and determine the cell count in sputum, as described below. In the latter phase of the study, the analytical results of sputum sample analysis requires that the researchers will be blinded to the classification of the sputum sample. To ensure sample adequacy as it relates to its collection for the deep lung, samples will be analyzed by a cytologist who will perform PAP staining for the presence of macrophages. Macrophages are an indication that the sputum sample is from deep within the lungs. Findings of the experiments and comparative study will not be used in the diagnosis or treatment of Participants.

Later optimization efforts including the comparative study will require that participants in the high-risk cohort undergo low dose computed tomography (LDCT) scans to confirm they do not have lung cancer. LDCT scans will be evaluated by a licensed, independent radiologist who may advise the participant to seek additional medical advice if warranted by LDCT imaging. Participants in the cancer cohort will have undergone LDCT scans identifying them as likely to have lung cancer prior to sample collection. Findings from the CyPath® Early Lung Cancer Detection Assay will not be used in the diagnosis of Participants or subsequent treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

* Male or female
* Study Participants must be willing to provide primary care physician contact information and agree to have medical information released if indicated
* Meet requirements of one of three cohorts in the study:

  * Healthy Cohort: Current non-smoker who has smoked less than 5 pack-years in his or her lifetime, and if smoked, has quit for more than 15 years ago and who has no known lung disease.
  * High Risk Cohort: Current smoker, or individual who has quit smoking less than 15 years before study start, who has smoked more than 30 pack-years in his or her lifetime.
  * Cancer Cohort: Individual who has been diagnosed by a physician with lung cancer.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

* Lung disease
* Angina with minimal exertion
* Pregnancy
* Have or have had cancer other than lung cancer
* Worked in the mining Industry

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 200 Participants will be recruited, 21 years of age or older of both sexes and all racial distributions. Participants must meet the exclusion criteria and inclusion criteria detailed under inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Assay Optimization | 320 days
  Assay optimization for methods to liquefy sputum by chemical dissociation, select proper fixatives and buffers, the efficacy of use of methyl-beta-cyclodextrin (MBCD) in sputum processing and determine the cell count in sputum. To ensure sample adequacy as deep lung, samples will be analyzed by a cytologist who will perform PAP staining for the presence of macrophages. Macrophages are an indication that the sputum sample is from deep within the lungs. Findings of the experiments and comparative study will not be used in the diagnosis or treatment of Participants.

SECONDARY OUTCOMES:
Identification of Differential Characteristics | 320 days
  Further optimization efforts including the comparative study will require that participants in the high-risk cohort undergo low dose computed tomography (LDCT) scans to confirm they do not have lung cancer. LDCT scans will be evaluated by a licensed, independent radiologist who may advise the participant to seek additional medical advice if warranted by LDCT imaging. Participants in the cancer cohort will have undergone LDCT scans identifying them as likely to have lung cancer prior to sample collection. Findings from the CyPath® Early Lung Cancer Detection Assay will not be used in the diagnosis of Participants or subsequent treatment decisions but provide comparative characteristics and correlation of sputum results between the three cohorts previously described between cohort samples and CyPath® Early Lung Cancer Detection Assay results

CONTACTS AND LOCATIONS:
Overall Officials: Vivienne Rebel, MD,PhD, Principal Investigator — bioAffinity Technologies
Locations (5):
- United States (5):
  - Waterbury Pulmonary Associates LLC, Waterbury, Connecticut
  - Meridian Health, Neptune City, New Jersey
  - Atlantic Respiratory Institute, Summit, New Jersey
  - Radiology Associates of Albuquerque, Albuquerque, New Mexico
  - bioAffinity Technologies, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patriquin L, Merrick DT, Hill D, Holcomb RG, Lemieux ME, Bennett G, Karia B, Rebel VI, Bauer T 2nd. Early Detection of Lung Cancer with Meso Tetra (4-Carboxyphenyl) Porphyrin-Labeled Sputum. J Thorac Oncol. 2015 Sep;10(9):1311-1318. doi: 10.1097/JTO.0000000000000627. PMID 26200451